CLINICAL TRIAL: NCT04762108
Title: Paediatric Sjögren Syndrome Cohort Study and Repository (PaedSSCoRe)
Acronym: PaedSSCoRe
Status: Active, not recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Children's Health Ireland (Other Government); Great Ormond Street Hospital (Unknown); Sheffield Children's NHS Foundation Trust (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 132557
Record Dates: First submitted 2021-02-15; First posted 2021-02-21 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Sjogren's Syndrome Childhood-onset
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood, tears, saliva, urine and glandular and extra-glandular (e.g. skin and renal) tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sjögren's syndrome: Sjögren's syndrome with childhood-onset
  Interventions: Other: Standard of care
- Healthy control: Age matched healthy control

INTERVENTIONS:
Other: Standard of care — Patients will be given standard of care as per their clinical needs
  Groups: Sjögren's syndrome

SUMMARY:
Sjögren syndrome (SS) in adults is characterised by inflammation of the exocrine glands, principally the salivary and lacrimal glands resulting in xerostomia (dry mouth) and xerophthalmia (dry eyes).It can also present with more extensive exocrinopathy as well as extra-glandular, systemic features.

SS is defined as primary SS (pSS) when it occurs in isolation, and as secondary SS, if associated with other autoimmune conditions. The incidence and prevalence rates of SS vary depending on the population. To date, there have been no studies reporting accurate incidence or prevalence of SS in childhood. Childhood onset SS defined as disease diagnosed before 18 years of age is believed to be rare; however, it is likely it is under-recognised and therefore under-diagnosed.

The overarching aim of this study is to identify epidemiological, clinical and laboratory characteristics of paediatric SS in a United Kingdom (UK) multi-centre cohort of patients. Using this data our goal is to develop universally accepted classification criteria that could be validated for use in a paediatric population.

Inclusion criterion for the study and repository is a diagnosis of SS made before 18 years by the referring physician. A data collection pack will be sent to authors willing to participate. Information collected will include but not exclusive to: demographic, clinical and laboratory/histological data at diagnosis and subsequent follow-up appointments. Biological samples including blood, tears, saliva, urine and glandular and extra-glandular (e.g. renal) tissue will be collected prospectively if available. Outcome measures related to disease activity and damage, as well as patient reported outcomes will also be collected at set time points (every 6 months) and during flares.

PaedSSCoRe will capture data on a significant cohort of children with SS providing a powerful resource to help improve our understanding of the pathogenesis and natural course of this disease.

Prospective data collection will allow a fuller analysis of poor prognostic features, impact of therapy and damage accrual, and variable outcome of childhood SS.

ELIGIBILITY:
Inclusion Criteria:

1. All recruited patients should be diagnosed with Sjogren's syndrome alone or in association with other autoimmune conditions (rheumatic or not) based on their rheumatologist opinion or have clinical and serological/imaging features which in the opinion of their clinician raise the suspicion of Sjogren's syndrome.
2. Patients with symptoms onset /imaging, serological and glandular biopsy abnormalities suggestive of SS (suspected SS) or SS diagnosis made by expert clinicians prior to age 18
3. Patients/ Carers who can provide informed consent and agree to provide access to the results of their routine care investigations for research purposes irrespective of being able provide blood or saliva samples.
4. Patients of 6 years or age or above

Exclusion Criteria:

1. Inability to provide informed consent or have informed consent provided on their behalf.

Min Age: 6 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Sjögren's syndrome with childhood-onset Healthy age matched controls Based on our preliminary estimations, there are currently 100-150 JSS patients under hospital care in the UK. The investigators envisaged to capture as many of the patients available, as well as the ones diagnosed for the duration of this project (10 years), estimating a recruitment number limit of 300 patients.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-01-11 (Actual); Primary Completion 2030-01-10 (Estimated); Study Completion 2030-01-10 (Estimated)

PRIMARY OUTCOMES:
Provide an estimate of the pre valence of relatively uncommon but serious manifestations of Sjögren's syndrome | 2 years
  Provide an estimate of the pre valence of relatively uncommon but serious manifestations of SS. The investigators will describe the prevalence of severe disease manifestations, such as lymphoma, central and peripheral nervous system and renal involvement (for which there is no data in paediatric populations) on all patients recruited to this cohort during this grant. The investigators will be correlating clinical manifestations to various parameters, such as age at onset, disease duration, ethnicity, gender, pubertal status, disease scores and patient and physician outcome measures aiming to establish disease trajectories.

SECONDARY OUTCOMES:
Explore immune signatures in a multi-centre cohort of childhood onset Sjögren's syndrome | 2 years
  The investigators aim to explore the specific immune signatures identified in adults in children and adolescent patients with paediatric onset SS. The investigators will assess their immune signatures (combined monocyte, B- and T-cell phenotype by multi-parameter flow cytometry)
Assess the metabolomic/transcriptomic profiles of paediatric Sjögren's syndrome endotypes | 2 years
  The pilot data from adults with SS suggest that certain endotypes could be enriched with an interferon-associated signature or metabolomic profile. Characterisation of these mechanisms could pinpoint additional novel biomarkers for endotype classification and potential novel targets for therapy.
Correlate -omic data with clinical and disease features to define the disease fingerprint associated with paediatric onset SS. | 2 years
  Following initial cleaning of data to remove metabolites/genes/cytokines showing no differences between paediatric SS patients and healthy donors, the investigators will stratify differentially expressed metabolic and genetic markers according to the identified immune-phenotypes and generate a disease fingerprint (combined -omics analysis) for paediatric SS. Correlations between gene expression and metabolomics and immune-phenotype (cells/cytokines) will be established using regression/cross-correlation analysis. The investigators will confirm which patterns of immune-phenotype/metabolic/ transcriptomic profiles are most highly associated with childhood-onset compared to adult SS endotypes.

CONTACTS AND LOCATIONS:
Locations (8):
- Children's Health Ireland (CHI) at Crumlin, Dublin, Ireland
- United Kingdom (7):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Great Ormond Street Hospital For Children NHS Foundation Trust, London
  - University College London Hospital, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Sheffield Children's NHS Foundation Trust, Sheffield
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No
The study will be complying to General Data Protection Regulation (GDPR) and Data protection regulations and personal identifiable information will not be made available to researchers under any circumstances. Data that will be shared will need to be approved by the steering committee in accordance to these regulations.